CLINICAL TRIAL: NCT05620628
Title: Ph2 Study of Savolitinib and Durvalumab (MEDI4736) Combination in Advanced MET Amplified Gastric Cancer(VIKTORY-2)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jeeyun Lee (Other)
Responsible Party: Sponsor-Investigator, Jeeyun Lee, Principal Investigator, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-06-110
Record Dates: First submitted 2022-11-03; First posted 2022-11-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Stomach Cancer, Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma | interventions — durvalumab; 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Savoritinib and Durvalumab (Experimental): A fixed dose of 1500 mg Q4W durvalumab (equivalent to 20 mg/kg Q4W) is used in the present study for patients >30 kg (dosing by bodyweight only required for patients ≤30 kg).And Savolitinib will be administered orally 600mg once a day for 28 days as one cycle.
  Interventions: Drug: Durvalumab; Drug: Savolitinib

INTERVENTIONS:
Drug: Durvalumab — Durvalumab will be administered at 1500mg every 4 weeks from cycles 1 day 1.
  Other Names: Imfinzi
Drug: Savolitinib — Savoritinib 600mg will be administered orally a day for 28 days as one cycle.
  Other Names: AZD6094

SUMMARY:
For patients who failed primary chemotherapy with MET amplification, The efficacy and safety of the chemotherapy are evaluated by using dervalumab and saboritinib in combination.

DETAILED DESCRIPTION:
Despite recent developments, the prognosis of patients with advanced gastric cancer is still poor, and the target treatment options studied in a recently completed randomized clinical trial in which patients with tumors expressing HER2 were treated with trastuzumab are proposed.

In this study, the survival period of patients treated with trastzumab was extended to less than 3 months. Despite these results, 80% of patients are still not eligible for trastzumab and need additional targeted therapy.

The largest somatic cell mutation frequency recorded in tumors can lead to higher renal antigen release and provision to the immune system. In addition, in some clinical trials, abnormal overexpression of MET was associated with poor clinical progress, rapid disease progression, and short survival period.

Double blocking of PD-1 and vascular endothelial growth factor receptor 2 appeared to increase inhibition of tumor growth compared to the treatment of each monoclonal antibody alone.

Therefore, in this study, the efficacy and safety of combination administration of immunoglobulin G1 that inhibits PD-L1 with MET amplification and Saboritinib (AZD6094), an MET inhibitor, are to be confirmed.

Histologically identified metastatic and recurrent gastric cancer, ECOG systemic activity of 0 or 1 and at least one measurable lesion in accordance with modified RECIST 1.1 According to the NGS results, the efficacy and safety of the combination administration of dervalumab and saboritinib are evaluated for gastric cancer patients scheduled for secondary and tertiary treatment with MET amplification.

Savoritinib is administered oral once a day at 600 mg (QD) every 28 days if it is more than 50 KG. Dervalumab is administered intravenously every four weeks from the first day of the first cycle CT will be used every 8 weeks from the first administration date to check the progress of the objective disease. Patients have evidence that they are resistant to treatment and useful in clinical trials, and if the supply of drugs is secured, they will continue to be treated with saboritinib and dervalumab.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥ 19 years of age
3. Body weight >30 kg
4. MET amplification by local NGS (The NGS result of the implementation agency is defined as copy number 4 or higher, which is the standard for amplification)
5. Patients with gastric cancer (GC) who are in progressive stages and have progressed during or after 1st or 2nd chemotherapy treatment, regardless of whether they are IO contactless (naïve) or IO
6. There shall be at least one measurable lesion according to the modified RECIST 1.1 criteria.
7. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
8. ECOG performance status 0-1 with no deterioration between screening and the first dose of study treatment
9. Patients must have a life expectancy ≥ 3 months from proposed first dose date.
10. Patients must have had a washout period of 2 weeks for any prior therapy prior to the start ot study drug. The following intervals between the end of the prior treatment and first dose of study drug must be observed: ≥ 4 weeks for radiotherapy (patients who receive palliative radiation for nontarget lesions need not have a 4 week washout period and can be enrolled if at least >=7 days); patients may receive a stable dose of bisphosphonates or denusomab as long as these were started at least 4 weeks prior to treatment; ≥ 4 weeks for major surgery; ≥ 7 days for minor surgical procedures; ≥ 14 days (or 5 half lives whoever is longest) for any investigational product.
11. Patients must have acceptable bone marrow, liver and renal function measured within 28 days prior to administration of study treatment as defined below:

    * Haemoglobin ≥9.0 g/dL (within 2 weeks of registration transfusion permitted)
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * Platelet count ≥100 x 109/L (within 2 weeks of registration transfusion permitted)
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x the upper limit of normal (ULN) with TBL≤ 1x ULN OR TBL >1ULN-≤1.5x ULN with ALT and AST ≤ 1x ULN
    * Serum creatinine ≤1.5 x institutional ULN
    * Glomerular filtration rate < 45 mL/min as assessed by standard methodology at the investigating centre
12. Female patients must be using highly effective contraception during clinical trials and for three months after permanent discontinuation of drug administration, and there should be evidence that they are not breastfeeding, that they are negative in pregnancy tests, or that they meet one of the following criteria in screening:
13. Male test subjects with a likely female spouse should be asked to use blocked contraception during the clinical trial and for six months after permanent cessation of administration of the test drug. The test subjects should avoid sperm donation from the start of the test treatment to the 6th month after permanent discontinuation.
14. optionally biopsy during the screening window prior to dosing and at progression (fresh frozen will be optionally if clinically feasible)

Exclusion Criteria:

1. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
2. Any previous treatment with MET inhibitors (prior exposure to anti-PD1/PDL1 allowed)<<if the study allows prior anti PD-1, PD-L1 and CTLA-4>> Patients who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4:
3. Any gastrointestinal condition that would preclude adequate absorption of savolitinib including but not limited to inability to swallow oral medication, refractory nausea and vomiting, chronic gastrointestinal diseases or previous significant bowel resection, intestinal obstruction or CTCAE grade 3 or grade 4 upper GI bleeding within 4 weeks before the enrollment.
4. Active or prior documented autoimmune or inflammatory disorders (including IBD[e.g. Chohn's disease, ulcerative colitis or diverticulitis], SLE, sarcoidosis syndrome, tuberculosis, Wegener syndrome, myasthenia gravis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, history of primary immunodeficiency.
5. Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
6. Active hepatitis B (positive HBV surface antigen (HBsAg) result) or hepatitis C (HCV).

   Patients with a past or resolved HBV infection are eligible if:
   * Negative for HBsAg and positive for hepatitis B core antibody [anti-HBcAb]. or:
   * Positive for HBsAg, but for > 6 months have had normal transaminases and HBV DNA levels <2000 IU/ml (ie, are in an inactive carrier state).
   * Subjects with HBV infection, characterised by positive HBsAg and/or anti-HBcAb with undetectable HBV DNA (< 10 IU/ml or under the limit of detection per local lab standard) do not require antiviral therapy prior to randomisation.

     * Patients with HBV infection, characterised by positive HBsAg and/or anti-HBcAb with detectable HBV DNA (≥ 10 IU/ml or above the limit of detection per local laboratory standard), must be treated with antiviral therapy for 2-4 weeks prior to the start of study treatment, with the choice of antivirals as per institutional practice. Following antiviral therapy initiation, subjects must show adequate viral suppression (ie, HBV DNA ≤ 2000 IU/mL) prior to randomisation. Participants will remain on antiviral therapy for the study duration and for at least 6 months after the last dose of IP Patients with positive HCV antibody are eligible only if the polymerase chain reaction is negative for HCV RNA.
7. Untreated central nervous system (CNS) metastatic disease, leptomeningeal disease, or cord compression. Note: Subjects previously treated for CNS metastases that are asymptomatic, radiographically and neurologically stable for at least 4 weeks and do not require corticosteroids (of any dose) for symptomatic management for at least 4 weeks prior to the first dose of treatment are not excluded.
8. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≤3 years.
9. Current or prior use of immunosuppressive medication within 4 weeks prior to the first dose of durvalumab, with the exceptions of intranasal, topical, and inhaled corticosteroids; systemic corticosteroids at physiologic doses not to exceed a dose > 10 mg prednisone / day or equivalent)
10. Patient was in receipt of any live attenuated vaccination within 30 days prior to study entry or within 30 days of receving study therapy.
11. Patients currently receiving (or unable to stop use at least 2 weeks) prior to receiving the first dose of savolitinib, medications known to be potent inhibitors of CYP1A2 or strong inducers of CYP3A4 with a narrow therapeutic range
12. Patient with any of the following cardiac criteria:

    -Mean QT interval corrected for heart rate (QTc) ≥ 470 ms calculated from 3 electrograms (ECGs) using Friderecia's correction . etc
13. Within 6months of treatment Any evidence of severe or uncontrolled systemic disease, including active infection (requiring antibiotics, antifungals or antivirals), diabetes type I and II, uncontrolled seizures, bleeding diatheses, severe COPD, severe Parkinson's disease.
14. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.

    For a unresolved toxicity,
15. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
16. Male or female patients who are familiar with pregnancy and contraception and have no intention of contraception.
17. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
18. History of allogenic organ transplantation.
19. Past history of PD-L1 or epileptic lung disease (ILD) or evidence of clinically active epileptic lung disease
20. History of liver cirrhosis of any origin and clinical stage; or history of other serious liver disease or chronic disease with relevant liver involvement, with or without normal LFTs*, such as Hemochromatosis,Alpha-1 Antitrypsin deficiency ,Autoimmune hepatitis (AIH), Primary sclerosing cholangitis (PSC), Primary biliary cirrhosis (PBC), Biopsy-confirmed Non-Alcoholic Steatohepatitis (NASH) with advanced fibrosis, Biopsy- confirmed Alcoholic Steatohepatitis with advanced fibrosis, Wilson's disease, Hepatocellular carcinoma

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
PFS (progression free survival) | up to 2years
  Efficacy of savolitinib combination with durvalumab

SECONDARY OUTCOMES:
ORR (objective response rate) | up to 2years
  Efficacy of savolitinib combination with durvalumab

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyun lee, Ph,MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No